CLINICAL TRIAL: NCT05938829
Title: Fetal Growth Restriction: Management Using Two Guidelines (FAME) - Fetal Growth Antenatal Management Evaluation
Brief Title: Fetal Growth Restriction: Management Using Two Guidelines - Fetal Growth Antenatal Management Evaluation
Acronym: FAME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Hector Mendez-Figueroa, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-2012
Record Dates: First submitted 2023-06-20; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-06

CONDITIONS: Fetal Growth Retardation
Keywords: antepartum surveillance
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasound using SMFM guidelines, then ultrasound using ISUOG guidelines (Other): Each site will utilize SMFM guidelines for the first 12 months and then there will be a 2 week washout period, after which each site will utilize ISUOG guidelines for 12 months
  Interventions: Other: Ultrasound following the SMFM guidelines; Other: Ultrasound following the ISUOG guidelines

INTERVENTIONS:
Other: Ultrasound following the SMFM guidelines — Patients will be followed with weekly ultrasound. During these scans, the patient will have a biophysical profile, a non-stress test (if the gestational age is over 32 weeks), and a Doppler interrogation of the fetal umbilical artery. This information will be captured in our ultrasound reporting software, Viewpoint.
Other: Ultrasound following the ISUOG guidelines — Patients will be followed with weekly ultrasound. During these scans, the patient will have a biophysical profile, a non-stress test (if the gestational age is over 32 weeks), and a Doppler interrogation of the fetal umbilical artery, middle cerebral artery, and ductus venosus. This information will be captured in our ultrasound reporting software, Viewpoint.

SUMMARY:
The purpose of this study is to compare the composite neonatal adverse outcomes (CNAO) among pregnancies complicated by fetal growth restriction (FGR) managed using the Society of Maternal-Fetal Medicine (SMFM) versus International Society of Ultrasound in Obstetrics and Gynecology (ISUOG) antepartum ultrasound guidelines, to measure the rate of the individual components of CNAO, to record the rate of cesarean delivery during labor, to tabulate the rate of deviation from the management protocol assigned at the time of evaluation, to record neonatal intensive care unit (NICU) admission rates and to measure the rate of the composite maternal adverse outcome (CMAO).

ELIGIBILITY:
Inclusion Criteria:

* FGR diagnosed during sonographic examinations
* estimated fetal weight less than or a fetal abdominal circumference less than the 10th percentile

Exclusion Criteria:

* Multiple gestations with FGR

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of neonates who have composite neonatal adverse outcomes (CNAO) | from time of birth to 30 days after birth

SECONDARY OUTCOMES:
Number of cesarean deliveries | at the time of delivery
Number of participants for whom there was a deviation from the management protocol | from time of diagnosis of fetal growth restriction to delivery
Number of participants that are admitted to neonatal intensive care unit (NICU) | from time of birth to 30 days after birth
Number of mothers who have composite maternal adverse outcomes (CMAO) | from time of birth to 30 days after birth
  This includes estimated blood loss (EBL) / quantitative blood loss (QBL) > 1,000 mL, Transfusion, chorioamnionitis, ICU admission, or Maternal death
Number of participants with Apgar score < 7 | at 5 minutes after birth
Number of participants that need mechanical ventilation | 6 hours after birth
Number of participants that show signs of neonatal seizure | from time of birth to 30 days after birth
Number of participants that have culture-proven neonatal sepsis | from time of birth to 30 days after birth
Number of participants that have intracranial hemorrhage | from time of birth to 30 days after birth
Number of participants that are still born or show neonatal death | from time of birth to 30 days after birth

CONTACTS AND LOCATIONS:
Overall Officials: Hector Mendez-Figueroa, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No